CLINICAL TRIAL: NCT05808335
Title: A Phase IIa Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Oral Antiviral Agents/hzVSF-v13 Combination Therapy vs Oral Antiviral Monotherapy in Chronic Hepatitis B Patients
Brief Title: A Study to Assess the Efficacy and Safety of Burfiralimab(hzVSF-v13) and OAD (Oral Antiviral Drug)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmuneMed, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM_hzVSF_v13-0003
Record Dates: First submitted 2023-03-27; First posted 2023-04-11 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo to hzVSF-v13 (Placebo Comparator): Placebo to match hzVSF-v13 + oral antiviral agent
  Interventions: Drug: Standard of care
- hzVSF-v13 50mg (Experimental): hzVSF-v13 50 mg/dose + oral antiviral agent
  Interventions: Drug: Standard of care
- hzVSF-v13 200mg (Experimental): hzVSF-v13 200 mg/dose + oral antiviral agent
  Interventions: Drug: Standard of care
- hzVSF-v13 800mg (Experimental): hzVSF-v13 800 mg/dose + oral antiviral agent
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Standard of care — The following medications listed are allowed to be administered during the course of the clinical study.
  1. Tenofovir (including salt-free or salt-modifying drugs)
  2. Entecavir (including salt-free or salt-modifying drugs)

SUMMARY:
This is a multicenter, randomized, double-blind, parallel group, 48-week follow-up, Phase IIa clinical study. This study has been designed to evaluate the change in HBsAg (log10 IU/mL) after administration of hzVSF-v13 50 mg/dose and hzVSF-v13 200 mg/dose in combination with an oral antiviral agent (Tenofovir or entecavir, including salt-free or salt-modifying drugs) compared to an oral antiviral agent in combination with a placebo (normal saline) in patients with chronic hepatitis B who are stably receiving an oral antiviral agent (Tenofovir or entecavir, including salt-free or salt-modifying drugs) for at least 24 weeks.

DETAILED DESCRIPTION:
Among the subjects who provided a voluntary written consent to participate in this clinical study, the patients with chronic hepatitis B who are stably receiving an oral antiviral agent (Tenofovir or entecavir, including salt-free or salt-modifying drugs) for at least 24 weeks prior to the screening visit can be considered as potential subjects of this study. Only the subjects who completed the final eligibility evaluation at the baseline visit (Visit 2) after the screening tests will be randomized to the hzVSF-v13 50 mg combination group, hzVSF-v13 200 mg combination group (study group) and placebo combination group (control group) at a 1:1:1 ratio at each site. The randomized subjects will receive intravenous administration of hzVSF-v13 or the placebo to match hzVSF-v13 four times with 4 weeks interval for a total of 12 weeks, and oral administration of 1 tablet of an oral antiviral agent will be given once daily for a total of 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Those who have a history of a diagnosis of chronic hepatitis B more than 24 weeks prior to screening and have been maintaining HBsAg positive at screening
2. Those who have an HBV DNA level that is below <20 IU/mL
3. Those who have been receiving tenofovir (including Tenofovir's salt-free or salt-modifying drugs), or entecarvir (including Entecavir's salt-free or salt-modifying drugs) stably for ≥24 weeks prior to screening and anticipated to maintain the identical drug with equivalent dosage and administration during the clinical trial.

Exclusion Criteria:

1. Those with a history of clinically significant chronic liver disease caused by other than chronic HBV infection at the time of screening
2. Patients with a signs of loss of liver function and decompensation of liver disease
3. Patients with uncontrolled diabetes (HbA1c >7.5%)
4. Patients with uncontrolled hypertension

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-03-27 (Estimated); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
Change in HBsAg from the baseline at 24 weeks (log10 IU/mL) | 24 weeks
  Baseline statistics for the changes in HBsAg (log10 IU/mL) from the baseline at 24 weeks shall be presented for each group, and a two-sample t-test or the Wilcoxon rank-sum test shall be performed to test differences of each study group compared to the control group.

SECONDARY OUTCOMES:
Percentage of subjects with HBsAg loss or seroconversion compared to the baseline at 8, 12, 24 and 48 weeks | 8, 12, 24, 48 weeks
  The number and percentage of subjects and 95% confidence interval for each treatment group and each evaluation time point shall be presented, and a chi-squared test or the Fisher's exact test shall be performed to test intergroup differences of each study group compared to the control group.
Percentage of subjects with HBV DNA lower than the lower limit of quantification (LLOQ) compared to the baseline at 24 and 48 weeks | 24, 48 weeks
  The number and percentage of subjects and 95% confidence interval for each treatment group and each evaluation time point shall be presented, and a chi-squared test or the Fisher's exact test shall be performed to test intergroup differences of each study group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Joon Hyeok Lee, M.D. Ph.D., Principal Investigator — Samsung Medical Center
Locations (4):
- South Korea (4):
  - Chung-Ang University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
It will be depending on internal discussion.